CLINICAL TRIAL: NCT05208580
Title: Impact of Patient Education on Preoperative Anxiety and Postoperative Psychosocial Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vilnius University (Other)
Collaborators: Vilnius University Hospital Santaros Klinikos (Other)
Responsible Party: Principal Investigator, Egle Kontrimaviciute, MD, PhD, Associate professor at Vilnius University, Lithuania, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/5-1351-823
Record Dates: First submitted 2021-10-03; First posted 2022-01-26 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Preoperative Anxiety

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- On-line education (Experimental): Virtual educational activities
  Interventions: Behavioral: Virtual education
- Contact education (Experimental): Live educational classes
  Interventions: Behavioral: Contact education
- Control group (No Intervention): Regular perioperative care without additional educational activities

INTERVENTIONS:
Behavioral: Virtual education — Participants undergo virtual education activities on an on-line platform 10-14 days before the surgery
  Arms: On-line education
Behavioral: Contact education — Participants attend live educational classes 10-14 days before the surgery
  Arms: Contact education

SUMMARY:
The aim of the study is to investigate the effect of preoperative patient education on the level of properative anxiety and postoperative psychosocial outcomes. Participants will be assigned to one of the 3 study groups: on-line education, contact education and control (no preoperative education). The investigators will evaluate preoperative anxiety level at different time points (baseline at 2 weeks before the surgery, at the evening before the surgery and postoperatively) and investigate dynamics of anxiety in the perioperative period. Additional qualitative interview by psychologists will be performed to evaluate the potential causes of increased/decreased preoperative anxiety.

Impact on postoperative complications, well-being of the participant, quality of recovery and satisfaction with medical care will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* agreement to participate in the study
* elective cholecystectomy or colon surgery

Exclusion Criteria:

* refusal to participate in the study
* do not speak Lithuanian
* do not pass the PHQ-2 depression screening test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-14 (Estimated)

PRIMARY OUTCOMES:
Change in preoperative anxiety level the day before the surgery in study groups | The day before the surgery
  Preoperative anxiety level will be compared with the baseline anxiety level evaluated at 10-14 days before the surgery. Anxiety level will be evaluated using Depression, Anxiety and Stress Scale 21 (DASS-21). Each of 21 item in a scale is evaluated using Likert-type scoring system (0 to 3 points, where 0 - not present, 3 - very consistent). The higher the socre, the higher the level of anxiety (worse outcome)
Change in preoperative anxiety and information level the day before the surgery in study groups | The day before the surgery
  Preoperative anxiety level will be compared with the baseline anxiety level evaluated at 10-14 days before the surgery. Anxiety and information levels will be evaluated using Amsterdam Preoperative Anxiety and Information Scale (APAIS). Scale consists of 6 questions (4 regarding anxiety and 2 regarding information about surgery and anesthesia). Each question is scored by five point Likert-type scale (1 to 5, where 1 - not at all, 5 - extremely). The higher the score, the higher the anxiety and need for information about surgery and anesthesia (worse outcome).

SECONDARY OUTCOMES:
Satisfaction with medical services | 48 hours after discharge from the hospital
  Evaluated using Hospital Consumer Assessment of Healthcare Providers and Systems questionnaire. Questionnaire consists of 29 questions about the recent hospital stay. Higher score - better satisfaction with medical care (better outcome).
Postoperative recovery | 48 hours after discharge from the hospital
  Evaluated using Quality of Recovery - 40 questionnaire. Questions are divided into part A and B. Each item in a questionnaire is evaluated by five point Likert-typescale (1 to 5, where 1 - never, 5 - all the time). Higher score accounts for more positive postoperative recovery process (better outcome).
Postoperative well-being of the patient | First 3 days of the postoperative period
  Subjective evaluation of well-being based on numerical scale 1 to 10 (1 - terrible, 10 - excellent) points. The higher the score, the better the outcome (postoperative well-being).
Postoperative pain levels | First 3 days of the postoperative period
  Evaluated using 11-point Numerical Pain Scale (0 - no pain, 10 - worst imaginable pain). Higher scores mean worse postoperative pain (worse outcome).
Postoperative delirium | First 3 days of the postoperative period
  Screening of delirium using Nursing Delirium Screening Scale. Includes 5 items, each is evaluated by 0 to 2 points. If the participant scores 2 points or more, the diagnosis of delirium is delivered.

OTHER OUTCOMES:
Causes of preoperative anxiety | Up to second postoperative week
  Qualitative interview performed by trained psychologists to evaluate potential causes of preoperative increased/decreased anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Egle Kontrimaviciute, MD, PhD, Principal Investigator — Vilnius University, Vilnius University Hospital Santaros Klinikos, Lithuania
Locations (1):
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided